CLINICAL TRIAL: NCT04824040
Title: Evaluation of Clinical, Immunological, Morphological, Molecular and Genetic Characteristics of Patients With Limb-girdle Muscular Dystrophy Type R2 (Type 2B) in the Russian Federation
Brief Title: Clinical, Immunological, Morphological and Genetic Characteristics of Patients With Dysferlinopathy (LGMD R2) in the RF
Acronym: DYSF-RUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Artgen Biotech (Other)
Collaborators: Genotarget (Industry)
Responsible Party: Sponsor
Other Study IDs: DYSF-Observation (RUS)
Record Dates: First submitted 2021-02-16; First posted 2021-04-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Dysferlinopathy; Miyoshi Myopathy; LGMDR2; DMAT
Keywords: LGMDR2; Miyoshi Myopathy; Dysferlinopathy; DYSF; DMAT
MeSH Terms: conditions — Dysferlinopathy; Miyoshi myopathy; Limb-girdle muscular dystrophy, type 2B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Patients with a genetically confirmed dysferlinopathy.
- Control group: Healthy Volunteers

SUMMARY:
To evaluate specific characteristics of phenotype, immune status, molecular and genetic as well as morphological characteristics of adult patients with limb-girdle muscular dystrophy R2 in various regions of the Russian Federation.

DETAILED DESCRIPTION:
A single-center, cohort clinical study. Subjects of both sexes aged 18 to 65 inclusive with genetically confirmed diagnosis of limb-girdle muscular dystrophy type R2, who have signed the written informed consent form for this study.

The control and case groups should be age- and gender-matched.

Study Objectives:

* To evaluate a clinical status of a subject (MMT score; 6-minute walk test; North Star Assessment for dysferlinopathy (NSAD));
* To assess blood biochemistry;
* To characterize muscle involvement based on MRI results;
* To evaluate the progression of muscle involvement based on repeated MRI;
* To assess cardiac function with ECG, EchoCG and MRI;
* To determine a gait pattern and balance characteristics in patients with limb-girdle muscular dystrophy using electrophysiological techniques (Neurosoft Gait Assessment System Steadys; stabilometrics and plantography with "SIDAS");
* To characterize changes in subpopulation compositions of T- and B-lymphocytes, phagocytic activity of leukocytes (a phagocytic index, a phagocyte number, an index of phagocytosis completeness, lysosomal-cation and NBT tests);
* To assess average blood cytokine levels in subjects with limb-girdle muscular dystrophy (type R2) in various regions of the Russian Federation;
* To assess average blood cytokine levels in healthy subjects from various regions of the RF;
* To analyze the relationship between blood cytokine levels and the presence of a mutation in the dysferlin gene;
* To study the expression (immunohistochemistry and western-blotting) and distribution of dysferlin in impaired muscles of subjects with LGMDR2.

The clinical study includes the stages as follows:

1. Subject enrollment - 24 months
2. Data collection and analysis - 12 months
3. Study Report - 30 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 (inclusive) years-old subjects of both sexes;
* A signed written informed consent form;
* Genetically confirmed diagnosis of limb-girdle muscular dystrophy (type 2B) (a case group)

Exclusion Criteria:

* A subject who is an investigator, study assistant, study coordinator and a member of the other personnel indirectly or directly associated with the conduct of the study;
* Acute medical conditions associated with visceral dysfunction, life-threatening conditions which occurred less than 6 months prior to enrollment into the study such as acute cardiac, renal, hepatic insufficiency, myocardial infarction or an acute cerebrovascular accident (stroke) as well as infectious diseases;
* Excessive alcohol consumption (> 20 g/day).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be identified through self-selection and direct recruitment options. Participants will be identified from the population of individuals who are followed at the neuromuscular clinics. Participants will also be solicited from the DYSF Russian registry.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Сlinical status of patients with dysferlinopathy (MMT score) | Through study completion at 24 months
  Muscle strength will be assessed using MMT and will be expressed in points for each of the muscle groups assessed.
Сlinical status of patients with dysferlinopathy ( North Star Assessment for dysferlinopathy) | Through study completion at 24 months
  North Star Assessment for Dysferlinopathy (NSAD) is a functional scale that will be used to measure motor performance in individuals with dysferlinopathy (includes 29 items).
Сlinical status of patients with dysferlinopathy (Hand Held Dynamometry). | Through study completion at 24 months
  Hand held dynamometry using the MicroFET2 myometer will be utilized to capture isometric muscle strength. Maximum strength in kilograms will be reported for each muscle group.
Сlinical status of patients with dysferlinopathy (6-minute walk test) | Through study completion at 24 months
  The participant will be asked to complete maximal distance in 6 minet as quickly as safely possible and the time in seconds is recorded.
Clinical blood test (level of hemoglobin) | Through study completion at 24 months.
  Level of hemoglobin is planned to be assessed in patients with dysferlinopathy.
Clinical blood test. Level of hematocrit | Through study completion at 24 months.
  Level of hematocrit (%) is planned to be assessed in patients with dysferlinopathy.
Clinical blood test. Level of RBC | Through study completion at 24 months.
  Level of RBC is planned to be assessed in patients with dysferlinopathy.
Clinical blood test. Level of WBC | Through study completion at 24 months.
  Level of WBC is planned to be assessed in patients with dysferlinopathy.
Clinical blood test. Levels of ESR | Through study completion at 24 months.
  Levels of ESR (mm/h) is planned to be assessed in patients with dysferlinopathy.
Clinical blood test. Level of platelets | Through study completion at 24 months.
  Level of platelets is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. | Through study completion at 24 months
  Levels of potassium (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of sodium | Through study completion at 24 months.
  Level of sodium (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of calcium | Through study completion at 24 months.
  Level of calcium (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of creatinine | Through study completion at 24 months.
  Level of creatinine (μmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of glucose | Through study completion at 24 months.
  Level of glucose (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of uric acid | Through study completion at 24 months.
  Level of uric acid (μmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of urea | Through study completion at 24 months.
  Level of urea (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of ALT | Through study completion at 24 months.
  Level of ALT (U/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of AST | Through study completion at 24 months.
  Level of AST (U/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of total protein | Through study completion at 24 months.
  Level of total protein (g/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of CPK | Through study completion at 24 months.
  Level of CPK (U/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of triglycerides | Through study completion at 24 months.
  Level of triglycerides (mmol/l) is planned to be assessed in patients with dysferlinopathy.
Biochemical blood test. Level of CRP | Through study completion at 24 months.
  Level of CRP (mg/l) is planned to be assessed in patients with dysferlinopathy.
Blood cytokine levels in subjects with dysferlinopathy and healthy volunteers. | Through study completion at 24 months
  * To assess average blood cytokine levels in subjects with dysferlinopathy in various regions of the Russian Federation;
  * To assess average blood cytokine levels in healthy subjects.
  Blood serum cytokine profiling will be performed with the use of the multiparameter fluorescent diagnostic system Luminex 200 and the Bio-Plex Pro Human 27-Plex Panel (Bio-Rad, Hercules, USA) in accordance with the manufacturer's instructions. The data obtained will be processed with the use of MasterPlex CT control and MasterPlex QT analysis software (Hitachi Software, San Bruno, USA).
  The following cytokine Levels will be assessed in the study:FGF2, Eotaxin,G-CSF, GM-CSF, IFN-γ, IL-1β, 1IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 p70, IL-13, IL-15, IL-17, IP-10, MCP-1/MCAF, MIP-1α, MIP-1β,PDGF-BB, RANTES, TNF-α, VEGF.
Autoantibodies in patients with dysferlinopathy. | Through study completion at 24 months
  Assessment of antibodу level against skeletal muscle antigens; an antinuclear factor (ANA), an extractable nuclear antigen.
Muscle MRI in patients with dysferlinopathy. | Through study completion at 24 months.
  * To characterize muscle involvement based on MRI results;
  * To evaluate the progression of muscle involvement based on repeated MRI once year;
Subpopulation compositions of T-lymphocytes in subjects with dysferlinopathy. | Through study completion at 24 months
  • To characterize changes in subpopulation compositions of T-lymphocytes in %.
Subpopulation compositions of B-lymphocytes in subjects with dysferlinopathy. | Through study completion at 24 months
  • To characterize changes in subpopulation compositions of B-lymphocytes in %.
Subpopulation compositions of phagocytic activity of leukocytes in subjects with dysferlinopathy (NBT test) | Through study completion at 24 months
  • To characterize changes in phagocytic activity of leukocytes (NBT test in CU).
Subpopulation compositions of phagocytic activity of leukocytes in subjects with dysferlinopathy. | Through study completion at 24 months
  • To characterize changes in phagocytic activity of leukocytes (a phagocyte number in CU).
Subpopulation compositions of phagocytic activity of leukocytes in subjects with dysferlinopathy (lysosomal-cation test). | Through study completion at 24 months
  • To characterize changes in phagocytic activity of leukocytes (lysosomal-cation test in CU).
Subpopulation compositions of phagocytic activity of leukocytes (a phagocytic index) in subjects with dysferlinopathy. | Through study completion at 24 months
  • To characterize changes in phagocytic activity of leukocytes (a phagocytic index).
Gait pattern and balance characteristics in patients with limb-girdle muscular dystrophy R2. | Through study completion at 24 months.
  To determine a gait pattern characteristics in patients with limb-girdle muscular dystrophy R2 using electrophysiological techniques (Neurosoft Gait Assessment System "STEDIS").
Cardiac function (assessed by Echocardiography). LV | Through study completion at 24 months.
  The absolute and relative sizes of the left ventricle (LV) index will be determined.
Cardiac function (assessed by Echocardiography). LV mass | Through study completion at 24 months.
  The absolute and relative sizes of the LV mass index will be determined.
Cardiac function (assessed by Echocardiography). Myocardium mass | Through study completion at 24 months.
  The absolute and relative sizes of the myocardium mass index will be determined.
Cardiac function (assessed by Echocardiography). RV | Through study completion at 24 months.
  The absolute and relative sizes of the right ventricle (RV) index will be determined.
Cardiac function (assessed by MRI scan with a gadolinium-based contrast agent). Volumetric evaluation of LV mass | Through study completion at 24 months.
  Volumetric evaluation of LV mass by manual tracing will be perform. An MRI of the heart will assess fibrosis.
Cardiac function (assessed by Echocardiography). LA | Through study completion at 24 months.
  The absolute and relative sizes of the left atrium (LA) index will be determined
Cardiac function (assessed by Electrocardiography). Outcome 13 | Through study completion at 24 months.
  To assess rhythm characteristic, P-wave, QRS, T-wave duration; PR, RR, QT intervals; PR, ST segments.
Cardiac function (assessed by MRI scan with a gadolinium-based contrast agent). Volumetric evaluation of EF | Through study completion at 24 months.
  Volumetric evaluation of EF by manual tracing will be performed.
Cardiac function (assessed by MRI scan with a gadolinium-based contrast agent). | Through study completion at 24 months.
  Volumetric evaluation of volume by manual tracing will be performed.
Morphological muscle study | Through study completion at 24 months.
  If it was necessary to confirm the causation of mutations in the dysferlin gene, the patients underwent muscle biopsy. To study the expression (immunohistochemistry and western-blotting) and distribution of dysferlin in impaired muscles of subjects with LGMDR2.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Deev, PhD, Study Chair — HSCI, Russia
Locations (1):
- Human Stem Cells Institute, Moscow, Russia

REFERENCES:
- [Background] Bardakov SN, Deev RV, Tsargush VA, Kaimonov VS, Musatova EV, Blagodatskikh KA, Tveleneva AA, Sofronova YV, Suslov VM, Carlier PG, Kurbatov SA, Yakovlev IA, Umakhanova ZR, Isaev AA. Asymptomatic and oligosymptomatic states of dysferlinopathy. J Neuromuscul Dis. 2024 Nov;11(6):1283-1294. doi: 10.1177/22143602241289227. Epub 2024 Dec 8. PMID 39973465
- [Background] Bardakov SN, Deev RV, Isaev capital A, Cyrilliccapital A, Cyrillic, Khromov-Borisov NN, Kopylov ED, Savchuk capital EM, CyrillicR, Pushkin MS, Presnyakov EV, Magomedova RM, Achmedova PG, Umakhanova ZR, Kaimonov VS, Musatova EV, Blagodatskikh Kcapital A, Cyrillic, Tveleneva Acapital A, Cyrillic, Sofronova YV, Yakovlev IA. Genetic screening of an endemic mutation in the DYSF gene in an isolated, mountainous population in the Republic of Dagestan. Mol Genet Genomic Med. 2023 Oct;11(10):e2236. doi: 10.1002/mgg3.2236. Epub 2023 Aug 8. PMID 37553796
- [Background] Umakhanova ZR, Bardakov SN, Mavlikeev MO, Chernova ON, Magomedova RM, Akhmedova PG, Yakovlev IA, Dalgatov GD, Fedotov VP, Isaev AA, Deev RV. Twenty-Year Clinical Progression of Dysferlinopathy in Patients from Dagestan. Front Neurol. 2017 Mar 8;8:77. doi: 10.3389/fneur.2017.00077. eCollection 2017. PMID 28337173
- [Background] Bardakov SN, Titova AA, Nikitin SS, Nikitins V, Sokolova MO, Tsargush VA, Yuhno EA, Vetrovoj OV, Carlier PG, Sofronova YV, Isaev capital A, Cyrilliccapital A, Cyrillic, Deev RV. Miyoshi myopathy associated with spine rigidity and multiple contractures: a case report. BMC Musculoskelet Disord. 2024 Feb 16;25(1):146. doi: 10.1186/s12891-024-07270-y. PMID 38365661
- [Background] Bardakov SN, Tsargush VA, Carlier PG, Nikitin SS, Kurbatov SA, Titova AA, Umakhanova ZR, Akhmedova PG, Magomedova RM, Zheleznyak IS, Emelyantsev AA, Berezhnaya EN, A Yakovlev I, Isaev AA, Deev RV. Magnetic resonance imaging pattern variability in dysferlinopathy. Acta Myol. 2021 Dec 31;40(4):158-171. doi: 10.36185/2532-1900-059. eCollection 2021 Dec. PMID 35047756
- [Background] Khaiboullina SF, Martynova EV, Bardakov SN, Mavlikeev MO, Yakovlev IA, Isaev AA, Deev RV, Rizvanov AA. Serum Cytokine Profile in a Patient Diagnosed with Dysferlinopathy. Case Rep Med. 2017;2017:3615354. doi: 10.1155/2017/3615354. Epub 2017 Apr 13. PMID 28487742